CLINICAL TRIAL: NCT00956930
Title: An Investigator Initiated Multicenter Prospective Randomized Study of Chemoembolization Versus Radioembolization for the Treatment of Hepatocellular Carcinoma (PREMIERE Trial)
Brief Title: Chemoembolization Versus Radioembolization in Treating Patients With Liver Cancer That Cannot Be Treated With Radiofrequency Ablation Or Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Riad Salem, Chief Vascular and Interventional Radiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 12339; P30CA060553 (NIH); STU# 00012339 (Other: Northwestern University IRB); CDR0000651416 (Other: PDQ)
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Liver Cancer
Keywords: advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (radioembolization) (Experimental): Patients undergo radioembolization with yttrium Y 90 glass microspheres by hepatic artery infusion for approximately 1-3 courses.
  Interventions: Radiation: yttrium Y 90 glass microspheres
- Arm II (transarterial chemoembolization [TACE]) (Experimental): Patients undergo TACE with mitomycin C, doxorubicin hydrochloride, and cisplatin by hepatic artery infusion for approximately 1-3 courses.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Radiation: yttrium Y 90 glass microspheres — Patients undergo radioembolization.
  Other Names: Radioembolization
  Arms: Arm I (radioembolization)
Drug: Doxorubicin — 75mg fixed dose
  Other Names: Doxorubicin hydrocholoride; Adriamycin; Chemoembolization (TACE)
  Arms: Arm II (transarterial chemoembolization [TACE])

SUMMARY:
RATIONALE: Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor. Radioembolization kills tumor cells by blocking the blood flow to the tumor and keeping radioactive substances near the tumor. It is not yet known which treatment regimen is more effective in treating patients with liver cancer.

PURPOSE: This randomized phase II trial is studying radioembolization to see how well it works compared with chemoembolization in treating patients with liver cancer that cannot be treated with Radiofrequency Ablation or removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare and contrast TACE and Y90 in order to determine either equivalence or superiority as measured by time-to-progression.

Secondary

* Characterize the safety and toxicity profile of these regimens.
* Determine the need for subsequent treatment in these patients.
* Determine tumor response in these patients
* Characterize change in quality of life and functional status in these patients.
* Determine time to progression in these patients.

OUTLINE: Patients are randomized to receive either TACE or Y90

* Arm I (radioembolization): Patients undergo radioembolization with yttrium Y 90 glass microspheres by hepatic artery infusion for approximately 1-3 courses.
* Arm II (transarterial chemoembolization [TACE]): Patients undergo TACE with mitomycin C, doxorubicin hydrochloride, and cisplatin by hepatic artery infusion for approximately 1-3 courses.
* In both arms, treatment modifications may apply according to response.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Hepatocellular Carcinoma confined to the liver that is unresectable with surgery or unable to be treated with radiofrequency ablation diagnosed by biopsy or imaging criteria (CT/MRI)
* No segmental, lobar, or main portal vein thrombosis as evidenced by CT or MRI imaging

Inclusion Criteria

* Adults > 18 years old of either gender
* Diagnosis of liver confined HCC confirmed by histology or American Association for the Study of Liver Diseases (AASLD) guidelines [59,60] [appendix A].
* Lesions < 1 cm in diameter have a low likelihood of being malignant and should be followed. Lack of growth over 1-2 years suggests it is not HCC.
* AFP >200 and radiological evidence (arterial hypervascularity) of lesion > 2 cm does not require biopsy.
* Two imaging modalities (triphasic CT, MRI, ultrasound, angiography) demonstrating "arterial hypervascularity" in the background of cirrhosis does not require biopsy
* One imaging modality with a lesion with arterial hypervascularity with wash out in early or delayed venous phase, does not require a biopsy
* Atypical appearances on imaging requires a biopsy.
* Non-conclusive biopsy requires closer monitoring
* For non-cirrhotics (by biopsy or imaging findings), diagnosis of HCC requires biopsy
* Patients with <50% liver involvement
* Measurable liver confined disease with bi-dimensional measurements, required within 4 weeks of screening. Lesions reported on imaging as "too small to characterize", abdominal lymph nodes < 2.0 cm or ascites in the setting of cirrhosis are not considered metastatic disease unless cytology proven.
* No segmental, lobar or main portal vein thrombosis as evidence by cross sectional imaging
* Prior resection permitted, no prior systemic, ablative or infusion therapy permitted
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 [appendix B]
* Childs score of A or B [appendix C]
* Required lab parameters within 28 days of screening
* Serum bilirubin ≤ 2.0 mg/dl (unless segmental infusion can be performed
* AST and ALT ≤ 5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Prothrombin time (PT)/ International normalized ratio (INR) ≤ 2.3 or PT ≤ 6 seconds above control. If subjects are being anticoagulated they can participate if proof of no coagulation abnormality existed prior to use of anticoagulants
* Negative serum or urine pregnancy test for females of child bearing potential
* Ability to understand and sign the informed consent; patient must have signed informed consent prior to registration on study
* Women of childbearing potential and sexually active males must use contraception while on study
* Lesions must be treatable angiographically by either radioembolization or chemoembolization.

Exclusion criteria

* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (angina symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Patients with infiltrative HCC are not eligible.
* Patients with bulk disease (≥70% tumor replacement of liver) are not eligible.
* Patients with ≥50% tumor replacement of liver, with an albumin < 3.0 g/dl are not eligible.
* Major surgery within 4 weeks prior to the screening visit
* Active clinically serious infection > Common Toxicity Criteria for Adverse Events (CTCAE v 4.0) Grade 2
* Any condition (psychological, physical or use/abuse of substances) which, in the opinion of the principal investigator (PI) or a sub-investigator (sub-I), would possibly endanger the subject during their participation in the study, or allow for non-compliance with the investigational drug and treatment under study.
* Due to the experimental nature of the therapy and the unknown risk to a fetus, pregnant and/or lactating women are not eligible to participate in this study.
* In the opinion of the investigator, patient is not a candidate/lesion not amenable for RFA (e.g. lesion location, shape, abnormal coagulation parameters, multi-focality).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2016-06-02 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published in medical journals.

REFERENCES:
- [Result] Salem R, Gordon AC, Mouli S, Hickey R, Kallini J, Gabr A, Mulcahy MF, Baker T, Abecassis M, Miller FH, Yaghmai V, Sato K, Desai K, Thornburg B, Benson AB, Rademaker A, Ganger D, Kulik L, Lewandowski RJ. Y90 Radioembolization Significantly Prolongs Time to Progression Compared With Chemoembolization in Patients With Hepatocellular Carcinoma. Gastroenterology. 2016 Dec;151(6):1155-1163.e2. doi: 10.1053/j.gastro.2016.08.029. Epub 2016 Aug 27. PMID 27575820
- See also: Y90 Radioembolization Significantly Prolongs Time to Progression Compared With Chemoembolization in Patients With Hepatocellular Carcinoma — https://www.ncbi.nlm.nih.gov/pubmed/27575820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All BCLC stage HCC patients were reviewed by the multidisciplinary tumor board(transplant surgery, hepatology, medical oncology, and interventional radiology) between October 2009 and October 2015.
Pre-assignment Details: 179 patients BCLC A/B patients were eligible. 43 declined to participate, 29 selected other clinical trials, 49 requested Y90 and 13 requested cTACE. 45 agreed to be randomized.
Period: Overall Study
Arm/Group | Arm I (Radioembolization) | Arm II (Transarterial Chemoembolization [TACE])
Started | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Radioembolization) | Arm II (Transarterial Chemoembolization [TACE]) | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: years] | 62 [58 to 65] | 64 [62 to 70] | 64 [58 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 19 | 16 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) in Patients Treated With TACE and Y90
Description: Compare and contrast TACE and Y90 in order to determine either equivalence or superiority as measured by time-to-progression. Patients have repeat imaging done (MRI or CT) at 1-month post procedure and then every 3 months after that. TTP and overall survival (OS) analyses were calculated from day of randomization by Kaplan-Meier analysis on intention-to-treat (ITT) basis.
  Progression (which is detected on follow-up imaging scans) was defined as:
  1. Progression by World Health Organization (WHO) response criteria 25% increase in bidimensional cross product.
  2. Progression by European Assosciation for the Study of the Liver (EASL): 25% increase in arterial enhancement
  3. Malignant portal vein tumor thrombus development
  4. Index lesion: lesions requiring re-treatment because of worsening circumferential enhancement
  5. Development of new lesions or extra-hepatic metastases.
Time Frame: Up to 6 yrs
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Radioembolization) | Arm II (Transarterial Chemoembolization [TACE])
Number analyzed (Participants) | 24 | 21
Months | 26 [14.5 to 26] | 6.8 [3.2 to 9.1]
Statistical Analysis 1: Comparison: Arm I (Radioembolization) vs Arm II (Transarterial Chemoembolization [TACE]); Test type: Superiority or Other; p = 0.007, Log Rank; Hazard Ratio (HR) = 0.122, 95% CI 2-sided [0.027 to 0.557]

2. Secondary Outcome: Number of Patients Who Achieved Complete or Partial Radiologic Response After Treatment
Description: Repeat imaging (CT/MRI) and lab work including tumor markers will be assessed 1 month post-treatment then every 3 months after that. Both EASL & WHO criteria are used.
  By EASL criteria Complete response is 100% Decrease in amount of enhancing tissue in index lesion, Partial response is ≥50% deecrease in amount of enhancing tissue in index lesion, Stable disease is <50% Decrease in to ≤ 25% increase in amount of enhancing tissue in index lesion, Progressive disease <25% Increase in amount of enhancing tissue in index lesion and/or new enhancement in previously treated index lesion.
Time Frame: up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Radioembolization) | Arm II (Transarterial Chemoembolization [TACE])
Number analyzed (Participants) | 23 | 19
Participants
  Complete & Partial Response Rate by EASL criteria | 20 | 14
  Stable Disease and progressive disease by EASL cri | 3 | 5

3. Secondary Outcome: Overall Survival
Description: Comparing overall survival of both treatment arms.
Time Frame: From day of randomization until date of death, or liver transplant or 7/15/2016, whichever came first, assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm I (Radioembolization): Patients undergo radioembolization with yttrium-90 glass microspheres by hepatic artery infusion for approximately 1-3 courses.
- Arm II (Transarterial Chemoembolization [TACE]): Patients undergo chemoembolization (TACE) with mitomycin C, doxorubicin hydrochloride, and cisplatin by hepatic artery infusion for approximately 1-3 courses.
  Doxorubicin: 75mg fixed dose
Arm/Group | Arm I (Radioembolization) | Arm II (Transarterial Chemoembolization [TACE])
Number analyzed (Participants) | 24 | 21
Months | 18.6 [7.4 to 32.5] | 17.7 [8.3 to 27.9]

ADVERSE EVENTS:
Time Frame: The study period included patients treated between October 2009 and June 2016. Patients were followed-up date of treatment up to date of last imaging, death or study closure, approximately 6 years
Description: Pts were followed up to date of last imaging, death, study closure (6 years). SAEs were reported if pts developed grade 3 or higher. Non SAEs reported if >1 pts developed grade 1-2. Two patients from arm II had follow-up at an outside hospital, both imaging and adverse-event related data were not available for us to include in the analyses. All efforts were made to obtain the data. Hence, they could not be included in the imaging/AE analysis. However, we were able to obtain survival status.
Arm/Group | Arm I (Radioembolization) | Arm II (Transarterial Chemoembolization [TACE])
All-Cause Mortality (participants affected / at risk) | 9/24 | 11/21
Serious Adverse Events (participants affected / at risk) | 6/24 | 3/19
Other Adverse Events (participants affected / at risk) | 24/24 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Radioembolization) (N=24) | Arm II (Transarterial Chemoembolization [TACE]) (N=19)
Abdominal Pain (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3 or 4 Abdominal Pain according to CTCAE V4.0
Fatigue (General disorders) | 0 (0) | 0 (0) — Grade 3 or 4 fatigue according to CTCAE (4.0)
Nausea (General disorders) | 0 (0) | 0 (0) — Grade 3 or 4 Nausea according to CTCAE (4.0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) — Grade 3 or 4 vomiting according to CTCAE (4.0)
Fever (General disorders) | 0 (0) | 0 (0) — Grade 3 or 4 fever according to CTCAE (4.0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) — Grade 3 or 4 anorexia according to CTCAE (4.0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) — Grade 3 or 4 constipation according to CTCAE (4.0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) — Grade 3 or 4 diarrhea according to CTCAE (4.0)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3 or 4 hypoalbuminemia according to CTCAE (4.0)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 1 (1) — Grade 3 or 4 bilirubin toxicity according to CTCAE (4.0)
Alkaline Phosphatase toxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) — Grade 3 or 4 alkaline phosphatase toxicity according to CTCAE (4.0)
Alanine aminotransferase toxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) — Grade 3 or 4 alanine aminotransferase toxicity according to CTCAE (4.0)
Aspartate aminotransferase toxicity (Hepatobiliary disorders) | 0 (0) | 2 (2) — Grade 3 or 4 aspartate aminotransferase toxicity according to CTCAE (4.0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 3 or 4 decrease in leukocyte count according to CTCAE (4.0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Grade 3 or 4 neutropenia according to CTCAE (4.0)
Liver Decompensation (Hepatobiliary disorders) | 3 (3) | 1 (1) — Hepatic function deterioration due to treatment or decompensation due to preexisting hepatic cirrhosis
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Infection of cutaneous and subcutaneous tissue
Hypokalemia (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 3 or higher hypokalemia
Sepsis (General disorders) | 2 (2) | 1 (1) — Development of severe generalized infection (sepsis).
OTHER ADVERSE EVENTS (reported when occurring in more than 0.04% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Radioembolization) (N=24) | Arm II (Transarterial Chemoembolization [TACE]) (N=19)
Fatigue (General disorders) | 21 (21) | 12 (12) — Grade 1 or 2 fatigue according to CTCAE (4.0)
Abdominal Pain (Hepatobiliary disorders) | 6 (6) | 10 (10) — Grade 1 or 2 abdominal pain according to CTCAE (4.0)
Nausea (General disorders) | 7 (7) | 8 (8) — Grade 1 or 2 nausea according to CTCAE (4.0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) — Grade 1 or 2 vomiting according to CTCAE (4.0)
Fever (General disorders) | 1 (1) | 3 (3) — Grade 1 or 2 fever according to CTCAE (4.0)
Anorexia (Gastrointestinal disorders) | 6 (6) | 4 (4) — Grade 1 or 2 anorexia according to CTCAE (4.0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1 or 2 Constipation according to CTCAE (4.0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) — Grade 1 or 2 diarrhea according to CTCAE (4.0)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1) | 11 (11) — Grade 1 or 2 hypoalbuminemia according to CTCAE (4.0)
Bilirubinemia (Hepatobiliary disorders) | 6 (6) | 5 (5) — Grade 1 or 2 hyperbilirubinemia according to CTCAE (4.0)
Alkaline Phosphatase toxicity (Hepatobiliary disorders) | 6 (6) | 2 (2) — Grade 1 or 2 alkaline Phosphatase toxicity according to CTCAE (4.0)
Alanine aminotransferase toxicity (Hepatobiliary disorders) | 3 (3) | 4 (4) — Grade 1 or 2 alanine aminotransferase toxicity according to CTCAE (4.0)
Aspartate aminotransferase toxicity (Hepatobiliary disorders) | 5 (5) | 7 (7) — Grade 1 or 2 aspartate aminotransferase toxicity according to CTCAE (4.0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — Grade 1 or 2 leukopenia according to CTCAE (4.0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 1 or 2 neutropenia according to CTCAE (4.0)

LIMITATIONS AND CAVEATS:
Limitations include small sample size and required censoring of imaging/survival to transplant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No